CLINICAL TRIAL: NCT02748187
Title: Are Therapist and Client Attachment Style and Reflective Functioning Associated With Outcomes in Cognitive Behavioural Analysis System of Psychotherapy (CBASP): A Longitudinal Proof of Concept Study
Brief Title: Attachment Style and Reflective Functioning in CBASP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15/SS/0232
Record Dates: First submitted 2016-03-27; First posted 2016-04-22 (Estimated); Last update posted 2024-05-03 (Actual); Status verified 2021-06

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Cognitive Behavioural Analysis System of Psychotherapy
  Interventions: Other: CBASP

INTERVENTIONS:
Other: CBASP — Interpersonal psychotherapy for chronic depression

SUMMARY:
Cognitive behavioural analysis system of psychotherapy (CBASP) is one of the only psychological models and treatments that has been designed specifically for patients diagnosed with chronic depression. CBASP in combination with antidepressants has been found to be the most effective treatment for chronic depression. Despite an increasing amount of research into this intervention, researchers are less aware of the role that specific and common ingredients are accounted for in outcomes. Given that CBASP is a treatment model endorsed by the National Health Service Scotland (NHS Scotland), gaining a deeper knowledge and understanding about the active ingredients involved in their success ensures current practice is embedded in an evidence base. Conducting this research adds to the gap in the literature and identifies areas in which further exploration is warranted. Given the emphasis on therapist variables in relation to treatment outcomes, the results of this research will have wider implications from a service resource perspective. Training may be altered or needs emphasised in line with the results of the study to ensure most efficacious outcomes.

Limited research has looked at therapist and client variables that may contribute to therapeutic alliance/engagement, and clinical outcomes. The current study proposes to explore two variables that are hypothesized to contribute to outcomes based on the theoretical framework CBASP is grounded on, namely therapist and client attachment style and reflective functioning. This will be done by providing CBASP to a small number of participants and gathering outcome data from therapists and clients at each therapy appointment. Participants will also complete the Adult Attachment Interview (AAI), a semi structured interview which can also be coded for reflective functioning. This is a proof of concept case series design that aims to provide an analysis of individual psychological change in relation to the above variables of interest.

DETAILED DESCRIPTION:
CBASP will consist of treatment of usual (i.e. one one-hour individual sessions on a weekly basis for up to 20 weeks) with additional outcome measures to be completed at each session. Therapists will receive a research pack which will outline when, and what, measures to administer and complete. To ensure anonymity and confidentiality of data collected, participants will be given identification numbers before data is submitted to a spread sheet for analysis.

9 CBASP therapists have been identified as suitable for participation in this study. Therapists will have the option to choose whether to take part in the research. Similarly, clients will be given the choice to take part in the research. To ensure at least one set of outcomes are achieved it is an aim of the study to provide the therapist with a minimum caseload of 2.

ELIGIBILITY:
Inclusion Criteria:

Clients will be included in this study if they meet the following criteria:

* Meet Diagnostic Statistical Manual-5 (DSM-5) criteria for persistent depressive disorder
* Have the capacity to provide informed consent
* Are aged 18 - 64 inclusive
* Speak fluent English
* Do not meet any of the exclusion criteria

Therapists will be included in the study if they meet the following criteria:

* Have received training in CBASP
* Have a qualification in at least one psychological therapy

Exclusion Criteria:

Clients will be excluded from the study if they do not meet inclusion criteria, as well as fulfilling any of the following criteria:

* Current significant substance misuse
* Undergoing other psychological treatment
* Presence of learning disability or significant cognitive impairment
* Presence of psychosis

Therapists will be excluded from the study if they do not meet the inclusion criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Psychological distress on the Clinical Outcome in Routine Evaluation Measure (CORE) | 5 minutes
  The CORE questionnaire, administered to clients, required 10 questions in relation to current mood to be answered. A total score is provided by adding up items. This is a routine outcome measure used in CBASP.
Depressive symptomology on the Patient Health Questionnaire (PHQ-9) | 5 minutes
  The PHQ-9 is a screening tool and monitor for depression that will be administered to clients. A total score is provided by adding up items.
Therapeutic relationship on the Working Alliance Inventory (WAI) | 10 minutes
  The WAI is a questionnaire that assesses the quality of the therapeutic relationship. There are two versions, namely client and therapist versions. Both therapists and clients will complete this questionnaire. A total score is provided by adding up items.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Buckley, BA, HDip, MA, Principal Investigator — University of Edinburgh
Locations (1):
- Sarah Buckley, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
via peer review journal

REFERENCES:
- [Result] Buckley; Attachment Style and Depression: An Investigation into Interpersonal Factors and Processes; DClinPsychol dissertation, available from https://era.ed.ac.uk/bitstream/handle/1842/25759/Buckley2017.pdf?sequence=1&isAllowed=y